CLINICAL TRIAL: NCT06539715
Title: Comparison of Visual Field Assessments Between Three Perimeters
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gainesville Eye Associates (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CB-24-01
Record Dates: First submitted 2024-07-25; First posted 2024-08-06 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- TEMPO (Experimental): Visual field assessment with the TEMPO
  Interventions: Diagnostic Test: Visual field assessment
- Humphrey Field Analyzer (Active Comparator): Visual field assessment with the Humphrey Field Analyzer
  Interventions: Diagnostic Test: Visual field assessment
- VisuALL (Active Comparator): Visual field assessment with the VisuALL
  Interventions: Diagnostic Test: Visual field assessment

INTERVENTIONS:
Diagnostic Test: Visual field assessment — Automated perimetry

SUMMARY:
A single center, prospective, randomized, comparative study of visual field assessments between the TEMPO, VisuALL, and HFA perimeters. Subjects will be assessed at 1 visit. Clinical evaluations will include MD, PSD, FT, VFI, OCT, and a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with best-corrected visual outcomes of 20/30 or better.

Exclusion Criteria:

* Unable to tolerate ophthalmic imaging
* Any ocular or systemic conditions, that could affect VF test results, such as age-related macular degeneration, peripheral retinal disease, or severe glaucoma.

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Total acquisition time (both eyes) | Visit 1 (Day 0)

SECONDARY OUTCOMES:
Mean deviation (MD) | Visit 1 (Day 0)
Pattern standard deviation (PSD) | Visit 1 (Day 0)
  PSD is a measure of visual field irregularity.
Foveal threshold (FT) | Visit 1 (Day 0)
  FT provides an estimate for best-corrected visual acuity.
Patient questionnaire | Visit 1 (Day 0)
  A series of 9 Likert style questions (Strongly Disagree to Strongly Agree) to assess comfort, ease of use, and anxiety with each device.

OTHER OUTCOMES:
Visual field index (VFI) | Visit 1 (Day 0)
Setup time | Visit 1 (Day 0)
False positives and false negatives (frequency) | Visit 1 (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Blehm, MD, Principal Investigator — North Georgia Eye Associates
Locations (1):
- North Georgia Eye Associates, Gainesville, Georgia, United States

IPD SHARING:
Plan to Share IPD: No